CLINICAL TRIAL: NCT01414517
Title: A Double-blind Placebo-controlled Trial of Dietary Supplementation With 15g/Day FOS for Five Weeks in Patients With Endometrial/Cervical Carcinoma or 7.5 Weeks in Patients With Prostate Carcinoma Undergoing Pelvic Radiotherapy.
Brief Title: Study to Prevent Radiation Induced Damage to Bowel Using a Prebiotic Enhanced Diet.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Responsible Party: Alastair Forbes Prof., University College London Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 09/H0715/61
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Radiation Enteritis; Radiation Proctitis
Keywords: Prebiotics; Acute Intestinal Injury; Chronic radiation enteritis
MeSH Terms: interventions — fructooligosaccharide; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOS (Active Comparator): Prebiotic (FructoOligoSaccharide-FOS.
  Interventions: Dietary Supplement: FructoOligoSaccharide
- Placebo (Placebo Comparator): Maltodextrin (non-prebiotic carbohydrate).
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: FructoOligoSaccharide — A mixture of 70% oligofructose and 30% inulin.
  Arms: FOS
Dietary Supplement: Maltodextrin — a non-prebiotic carbohydrate
  Arms: Placebo

SUMMARY:
The study will consist of pair of double-blind placebo-controlled trials of dietary supplementation with 15g/day FructoOligoSaccharide (FOS) for 7.5 weeks in patients with prostate carcinoma or 5 weeks in patients with cervical or endometrial carcinoma who are to undergo pelvic radiotherapy with intent to cure.

DETAILED DESCRIPTION:
The study will consist of pair of double-blind placebo-controlled trials of dietary supplementation with 15g/day FructoOligoSaccharide (FOS) for 7.5 weeks in patients with prostate carcinoma or 5 weeks in patients with cervical/endometrial carcinoma who are to undergo pelvic radiotherapy with intent to cure. Patients having post-operative adjuvant irradiation will be eligible, but not those having purely palliative treatment for symptom control. The clinical trials will be based at University College Hospital. Patients will attend a screening visit, a baseline visit, and follow-up visits at completion of radiotherapy, and then at three and six months.

Patients will be randomised to take a daily dietary supplement of either placebo (a non-prebiotic carbohydrate) or FOS (a mixture of 70% oligofructose and 30% inulin), provided as a single 15g sachet that can be dissolved in water or added to food. Randomisation in the gynaecological trial will be stratified according to diagnosis. In other respects management will be that offered routinely to patients undergoing pelvic radiotherapy for prostate malignancy or endometrial/cervical malignancy.

The studies are powered to detect the primary outcome measure of a clinical response (lower frequency of acute radiation enteritis/proctitis at 5 or 7.5 weeks respectively) using a 2-sample binomial arcsine where the predicted rate of acute radiation induced bowel disease when on FOS is 50% and 80% on placebo, to a significance of 0.05 and at a power of 90%.

Fifty-one patients will be required in each group to detect a significant difference between FOS and placebo. Therefore 110 patients will be recruited to each of the two studies to allow for attrition.

The primary endpoint will be the clinical gastrointestinal status at 7.5 weeks or 5 weeks at completion of radiotherapy. This status will be enumerated in comparison with placebo treated patients from the Birmingham score of intestinal symptoms (a simple clinical score from 0-15, usually employed in ulcerative colitis). Most patients commencing radiotherapy for these malignancies will have a pre-treatment score of zero or 1. A score of 4 or more is indicative of active coloproctitis, and differences of more than 2 points are to be considered clinically meaningful.

Secondary clinical endpoints will include the quantity of anti-diarrhoeal medication required, the international harmonised criteria for radiation toxicity, the EuroQol score of quality of life, and the appearance of the rectal mucosa: as judged endoscopically using the Baron score (a 0-3 scale usually employed in ulcerative colitis); and semi-quantitatively from histological assessment.

The Birmingham score and each of the clinical secondary endpoints will be assessed again at 3 and 6 months after completion of the radiotherapy. Endoscopic and histological assessment will be repeated only at 6 months after completion of radiotherapy.

Laboratory endpoints will include the measurement of short chain fatty acids (SCFA) (including butyrate) in faeces at baseline and at completion of radiotherapy, and study of the microbiota profile in the mucosa as determined by fluorescence in-situ hybridization (FISH). Haematological and biochemical parameters will be monitored as in standard practice.

ELIGIBILITY:
Inclusion Criteria:

* The study group will comprise men and women aged 18 years or older with a histologically proven diagnosis of carcinoma of the prostate or carcinoma of the cervix or endometrium in whom radical radiotherapy has been selected in their treatment plan following assessment by the prostate oncology or gynecological oncology multidisciplinary team

Exclusion Criteria:

* Exclusion criteria will preclude the recruitment of those having radiotherapy for purely palliative reasons. Patients known to have a current infection with an enteric pathogen, or who have used antibiotics within the past month, consumed any probiotic or prebiotic within the last month, or used any rectal/topical therapy within the last month will also be ineligible. Those known or suspected to have inflammatory bowel disease (ulcerative colitis or Crohn's disease) will be ineligible. Patients requiring hospitalisation, and those considered by the chief investigator (CI) to have important hepatic, renal, endocrine, respiratory, neurological or cardiovascular disease will also be ineligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-06 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Status | 5 weeks or 7.5 weeks
  To determine whether there is a difference in gastrointestinal status at 5 weeks (enumerated through the Birmingham score) in patients undergoing pelvic irradiation for gynaecological malignancy or at 7.5 weeks in patients undergoing radiotherapy for prostate malignancy given a prebiotic enhanced diet and those on placebo.

SECONDARY OUTCOMES:
Short Term Toxicity | 5 weeks or 7.5 weeks
  To determine the effects of FOS on the short-term toxicity of pelvic irradiation (in comparison to placebo).
See Effects of FOS | 5 or 7.5 weeks, 6 months
  To establish the effects of FOS on intestinal integrity, determined endoscopically, biochemically and histologically, after pelvic irradiation, both immediately and at 6 months follow-up
Effect of FOS on Chronic Radiation Bowel Disease | 5 weeks or 7.5 weeks, 3 months, 6 months
  To provide pilot data to determine whether FOS given during pelvic irradiation has an effect on the risk of clinically apparent chronic radiation bowel disease.
Effect on Gut Microbiota | 5 weeks or 7.5 weeks, 3 months, 6 months
  To confirm using fluorescence in-situ hybridization (FISH) the changes in the gut microbiota in patients on FOS enhanced diet in comparison with standard diet.

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Forbes, Bsc;MD;FRCP;FHEA, Principal Investigator — University College London Hospitals/University College London
Locations (1):
- University College London Hospital, London, London, United Kingdom